CLINICAL TRIAL: NCT04589845
Title: Tumor-agnostic Precision Immuno-oncology and Somatic Targeting Rational for You (TAPISTRY) Phase II Platform Trial
Brief Title: Tumor-agnostic Precision Immuno-oncology and Somatic Targeting Rational for You (TAPISTRY) Platform Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO41932; 2020-001847-16 (EudraCT Number); 2023-507418-28-00 (EU CTIS Number)
Record Dates: First submitted 2020-10-11; First posted 2020-10-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors
MeSH Terms: interventions — entrectinib; alectinib; atezolizumab; ipatasertib; Ado-Trastuzumab Emtansine; inavolisib; pralsetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Cohort A: ROS Proto-oncogene 1 (ROS1) Fusion-positive Tumors (Excluding NSCLC) (Experimental): Participants with metastatic or advanced solid tumors, with the exception of non-small cell lung cancer (NSCLC), will receive entrectinib once daily (QD) in repeated 28-day cycles at a dose of 600 milligram per day (mg/day) for adults and pediatric participants with a body surface area (BSA) ≥ 1.51 square meter (m^2). The total dose of daily entrectinib administration for pediatric participants with BSA < 1.51 m^2 will be lower.
  Interventions: Drug: Entrectinib
- Cohort B: Neurotrophic Tyrosine Receptor Kinase (NTRK) 1/2/3 Fusion-positive Tumors (Experimental): Participants with metastatic or advanced solid tumors will receive entrectinib, QD in repeated 28-day cycles at a dose of 600 mg/day for adults and pediatric participants with a BSA ≥ 1.51 m^2. The total dose of daily entrectinib administration for pediatric participants with BSA < 1.51 m^2 will be lower.
  Interventions: Drug: Entrectinib
- Cohort C: Anaplastic Lymphoma Kinase (ALK) Fusion-positive Tumors (Excluding NSCLC) (Experimental): Participants with metastatic or advanced solid tumors, with the exception of NSCLC, will receive alectinib at a dosage of 600 mg, orally, twice a day (BID), taken with food, in repeated 28-day cycles.
  Interventions: Drug: Alectinib
- Cohort D: TMB-high Tumors (Experimental): Participants with metastatic or advanced solid tumors will receive atezolizumab intravenously (IV) at a fixed dose for participants aged ≥ 18 years, and 15 milligrams per kilogram (mg/kg) (maximum 1200 mg) for participants aged < 18 years on Day 1 of each 21-day cycle. Note: Cohort D has been closed for enrollment.
  Interventions: Drug: Atezolizumab
- Cohort E: Protein Kinase B (AKT) 1/2/3 Mutant-positive Tumors (Experimental): Participants with metastatic or advanced solid tumors will receive ipatasertib orally, QD at the starting dose of 400 mg in repeated 28-day cycles until the participant experiences disease progression, intolerable toxicity, or withdraws consent. For participants 12-17 years of age, ipatasertib will be administered at the starting dose of 200 mg for participants < 35 kilograms (kg), 300 mg for participants ≥ 35 and < 45 kg, 400 mg for those ≥ 45 kg orally QD in repeated 28-day cycles until the participant experiences disease progression, intolerable toxicity, or withdraws consent. Note: Cohort E has been closed for enrollment.
  Interventions: Drug: Ipatasertib
- Cohort F: Human Epidermal Growth Factor Receptor 2 (HER2) Mutant-positive Tumors (Experimental): Participants with metastatic or advanced solid tumors will receive trastuzumab emtansine IV at a dose of 3.6 mg/kg every 21 days.
  Note: Cohort F has been closed as of protocol version 7 because enrollment and participant follow-up have been completed.
  Interventions: Drug: Trastuzumab emtansine
- Cohort H: PIK3CA Multiple Mutant-positive Tumors (Experimental): Participants with phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA) multiple mutant-positive tumors will receive inavolisib (GDC-0077) QD at a starting dose of 9 mg by mouth (PO) in repeated 28-day cycles. Note: Cohort H has been closed for enrollment.
  Interventions: Drug: Inavolisib
- Cohort I: BRAF Class II Mutant or Fusion-positive Tumors (Experimental): Participants with proto-oncogene B-Raf (BRAF) class II mutant/fusion-positive tumors (adults and adolescents ≥ 40 kg) will receive 400 mg belvarafenib, PO, BID with adequate water (more than 200 milliliters [mL]). One cycle consists of 28 days. Administration of belvarafenib should occur BID on every day of each 28-day cycle. Note: Cohort I has been closed for enrollment.
  Interventions: Drug: Belvarafenib
- Cohort J: BRAF Class III Mutant-positive Tumors (Experimental): Participants with BRAF class III mutant-positive tumors (adults and adolescents ≥ 40 kg) will receive 400 mg belvarafenib PO BID with adequate water (more than 200 mL). One cycle consists of 28 days. Administration of belvarafenib should occur BID on every day of each 28-day cycle. Note: Cohort J has been closed for enrollment.
  Interventions: Drug: Belvarafenib
- Cohort K: Rearranged During Transfection (RET) Fusion-positive Tumors (Excluding NSCLC) (Experimental): Participants with RET fusion-positive tumors will self-administer pralsetinib orally at home (except on clinic days) on a continuous daily dosing regimen at a dose of 400 mg/day (four 100-mg capsules per day) for adult and pediatric participants ≥ 12 and < 18 years of age. A treatment cycle consists of 4 weeks (28 days). Note: Cohort K has been closed for enrollment.
  Interventions: Drug: Pralsetinib
- Cohort L: KRAS G12C-positive Tumors (Excluding NSCLC and Colorectal Cancer [CRC]) (Experimental): Participants with kirsten rat sarcoma virus (KRAS) G12C-positive tumors will self-administer divarasib (GDC-6036) orally at home (except on clinic days).
  Interventions: Drug: Divarasib
- Cohort M: Ataxia-telangiectasia Mutated (ATM) Loss of Function (LOF) Tumors (Experimental): Participants with ATM LOF tumors will self-administer camonsertib orally at home (except on clinic days).
  Interventions: Drug: Camonsertib
- Cohort N: SETD2 LOF Tumors (Experimental): Participants with methyltransferase SET (Su(var) 3-9) Enhancer of zest and Trithorax) domain-containing 2 (SETD2) LOF tumors will self-administer camonsertib orally at home (except on clinic days).
  Interventions: Drug: Camonsertib

INTERVENTIONS:
Drug: Entrectinib — Adults and pediatric participants with a BSA ≥1.51 m^2: entrectinib will be self-administered by participants orally at home at a dose of 600 mg/day (three 200-mg capsules per day). Pediatric participants with a BSA < 1.51 m^2: entrectinib will be administered orally at home in mini-tablet formulation at a dose of 400 mg/day (BSA=1.11-1.50 m^2) or 300 mg/day (BSA=0.81-1.10 m^2) or 200 mg/day (BSA=0.51-0.80 m^2) or 300 milligrams per square meter (mg/m^2) (BSA=0.43-0.50 m^2).
  Other Names: Rozlytrek
  Arms: Cohort A: ROS Proto-oncogene 1 (ROS1) Fusion-positive Tumors (Excluding NSCLC)
Drug: Entrectinib — Adults and pediatric participants with a BSA ≥ 1.51 m^2: entrectinib will be self-administered by participants orally at home at a dose of 600 mg/day (three 200-mg capsules per day). Pediatric participants with a BSA < 1.51 m^2: entrectinib will be administered orally at home in mini-tablet formulation at a dose of 400 mg/day (BSA=1.11-1.50 m^2) or 300 mg/day (BSA=0.81-1.10 m^2) or 200 mg/day (BSA=0.51-0.80 m^2) or 300 mg/m^2 (BSA=≤0.50 m^2).
  Other Names: Rozlytrek
  Arms: Cohort B: Neurotrophic Tyrosine Receptor Kinase (NTRK) 1/2/3 Fusion-positive Tumors
Drug: Alectinib — Alectinib will be administered orally BID with food at a dosage of 600 mg (four 150-mg capsules).
  Other Names: Alecensa
  Arms: Cohort C: Anaplastic Lymphoma Kinase (ALK) Fusion-positive Tumors (Excluding NSCLC)
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at a fixed dose of 1200 mg for participants aged ≥18 years, and 15 mg/kg (maximum 1200 mg) for participants aged <18 years on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
  Arms: Cohort D: TMB-high Tumors
Drug: Ipatasertib — For participants 12-17 years of age, ipatasertib will be administered at the starting dose of 200 mg for participants < 35 kg, 300 mg for participants ≥35 and < 45 kg, 400 mg for those ≥ 45 kg orally QD, beginning of Cycle 1, on Days 1-21 of each 28-day cycle until the participant experiences disease progression, intolerable toxicity, or withdraws consent.
  Arms: Cohort E: Protein Kinase B (AKT) 1/2/3 Mutant-positive Tumors
Drug: Trastuzumab emtansine — Trastuzumab emtansine will be administered at 3.6 mg/kg by IV infusion every 21 days until disease progression or unacceptable toxicity. The dosage and administration method also applies for pediatric participants 12-17 years of age.
  Other Names: Kadcyla
  Arms: Cohort F: Human Epidermal Growth Factor Receptor 2 (HER2) Mutant-positive Tumors
Drug: Inavolisib — GDC-077 will be administered QD at a starting dose of 9 mg PO in repeated 28-day cycles. The dosage and administration method also applies for pediatric participants 12-17 years of age.
  Other Names: GDC-0077
  Arms: Cohort H: PIK3CA Multiple Mutant-positive Tumors
Drug: Belvarafenib — Belvarafenib will be administered at a dose 400 mg, PO, BID with adequate water (more than 200 mL). One cycle consists of 28 days. Administration of belvarafenib should occur BID on every day of each 28-day cycle.
  Arms: Cohort I: BRAF Class II Mutant or Fusion-positive Tumors; Cohort J: BRAF Class III Mutant-positive Tumors
Drug: Pralsetinib — Pralsetinib will be self-administered by participants orally at home (except on clinic days) on a continuous daily dosing regimen at a dose of 400 mg/day (four 100-mg capsules per day) for adult and pediatric participants ≥ 12 and < 18 years of age. A treatment cycle consists of 4 weeks (28 days).
  Other Names: Gavreto (US)
  Arms: Cohort K: Rearranged During Transfection (RET) Fusion-positive Tumors (Excluding NSCLC)
Drug: Divarasib — Divarasib will be self-administered by participants orally at home (except on clinic days) on a continuous daily dosing regimen for both adult and pediatric participants. A treatment cycle consists of 3 weeks (21 days).
  Other Names: GDC-6036
  Arms: Cohort L: KRAS G12C-positive Tumors (Excluding NSCLC and Colorectal Cancer [CRC])
Drug: Camonsertib — Camonsertib will be self-administered by participants orally at home (except on clinic days). A treatment cycle consists of 3 weeks and will be given on days 1-3 and days 8-10 of every 21-day cycle.
  Arms: Cohort M: Ataxia-telangiectasia Mutated (ATM) Loss of Function (LOF) Tumors; Cohort N: SETD2 LOF Tumors

SUMMARY:
TAPISTRY is a Phase II, global, multicenter, open-label, multi-cohort study designed to evaluate the safety and efficacy of targeted therapies or immunotherapy as single agents or in rational, specified combinations in participants with unresectable, locally advanced or metastatic solid tumors determined to harbor specific oncogenic genomic alterations or who are tumor mutational burden (TMB)-high as identified by a validated next-generation sequencing (NGS) assay. Participants with solid tumors will be treated with a drug or drug regimen tailored to their NGS assay results at screening. Participants will be assigned to the appropriate cohort based on their genetic alteration(s). Treatment will be assigned on the basis of relevant oncogenotype, will have cohort-specific inclusion/exclusion criteria, and, unless otherwise specified, will continue until disease progression, loss of clinical benefit, unacceptable toxicity, participant or physician decision to discontinue, or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced and unresectable or metastatic solid malignancy
* Measurable disease as defined by RECIST v1.1, RANO, or INRC
* Performance status as follows: Participants aged ≥ 18 years: Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2; Participants aged 16 to < 18 years: Karnofsky score ≥ 50%; Participants aged < 16 years: Lansky score ≥ 50%
* For participants aged ≥ 18 and < 18 years: adequate hematologic and end-organ function
* Disease progression on prior treatment, or previously untreated disease with no available acceptable treatment
* Adequate recovery from most recent systemic or local treatment for cancer
* Life expectancy ≥ 8 weeks
* Ability to comply with the study protocol, in the investigator's judgment
* For female participants of childbearing potential: Negative serum pregnancy test ≤ 14 days prior to initiating study treatment, agreement to remain abstinent or use single or combined contraception methods that result in a failure rate of < 1% per year for the period defined in the cohort-specific inclusion criteria; and agreement to refrain from donating eggs during the same period
* For male participants: Willingness to remain abstinent or use acceptable methods of contraception as defined in the cohort-specific inclusion criteria
* In addition to the general inclusion criteria above, participants must meet all of the cohort-specific inclusion criteria for the respective cohort

Exclusion Criteria:

* Current participation or enrollment in another therapeutic clinical trial
* Any anticancer treatment within 2 weeks or 5 half-lives prior to start of study treatment
* Whole brain radiotherapy within 14 days prior to start of study treatment
* Stereotactic radiosurgery within 7 days prior to start of study treatment
* Pregnant or breastfeeding, or intending to become pregnant during the study
* History of or concurrent serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study or confounds the ability to interpret data from the study
* Incomplete recovery from any surgery prior to the start of study treatment that would interfere with the determination of safety or efficacy of study treatment
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or higher), myocardial infarction, or cerebrovascular accident within 3 months prior to enrollment, unstable arrhythmias, or unstable angina
* History of another active cancer within 5 years prior to screening that may interfere with the determination of safety or efficacy of study treatment with respect to the qualifying solid tumor malignancy
* In addition to the general exclusion criteria above, in order to be enrolled in a treatment cohort of the study, participants must not meet any of the cohort-specific exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 920 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2032-09-25 (Estimated); Study Completion 2032-09-25 (Estimated)

PRIMARY OUTCOMES:
All Cohorts: Independent Review Committee (IRC)-assessed Objective Response Rate (ORR) Based on Confirmed Objective Response (OR) per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Approximately up to 12 years
  Confirmed objective response indicates ≥4 weeks after initial documentation of response.

SECONDARY OUTCOMES:
All Cohorts: IRC-assessed Duration of Response (DOR) per RECIST v1.1 | Approximately up to 12 years
All Cohorts: IRC-assessed Clinical Benefit Rate (CBR) per RECIST v1.1 | Approximately up to 12 years
All Cohorts: IRC-assessed Progression-free Survival (PFS) per RECIST v1.1 | Approximately up to 12 years
All Cohorts: Investigator (INV)-assessed ORR per RECIST v1.1 | Approximately up to 12 years
All Cohorts: INV-assessed DOR per RECIST v1.1 | Approximately up to 12 years
All Cohorts: INV-assessed CBR per RECIST v1.1 | Approximately up to 12 years
All Cohorts: INV-assessed PFS per RECIST v1.1 | Approximately up to 12 years
All Cohorts: IRC- and INV-assessed Time to Central Nervous System (CNS) Progression per RECIST v1.1 | Approximately up to 12 years
All Cohorts: Overall Survival (OS) | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: IRC-assessed CNS-ORR per Response Assessment in Neuro-oncology (RANO) | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: IRC-assessed CNS-DOR per RANO | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: IRC-assessed CNS-CBR per RANO | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: IRC-assessed CNS-PFS per RANO | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: INV-assessed CNS-ORR per RANO | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: INV-assessed CNS-DOR per RANO | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: INV-assessed CNS-CBR per RANO | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: INV-assessed CNS-PFS per RANO | Approximately up to 12 years
Cohorts A, B, C, D, E, F, H, I, J, K, L, M, N: IRC-assessed ORR per International Neuroblastoma Response Criteria (INRC) | Approximately up to 12 years
Cohorts A, B, C, D, E, F, H, I, J, K, L, M, N: IRC-assessed DOR per INRC | Approximately up to 12 years
Cohorts A, B, C, D, E, F, H, I, J, K, L, M, N: IRC-assessed CBR per INRC | Approximately up to 12 years
Cohorts A, B, C, D, E, F, H, I, J, K, L, M, N: IRC-assessed PFS per INRC | Approximately up to 12 years
Cohorts A, B, C, D, E, F, H, I, J, K, L, M, N: INV-assessed ORR per INRC | Approximately up to 12 years
Cohorts A, B, C, D, E, F, H, I, J, K, L, M, N: INV-assessed DOR per INRC | Approximately up to 12 years
Cohorts A, B, C, D, E, F, H, I, J, K, L, M, N: INV-assessed CBR per INRC | Approximately up to 12 years
Cohorts A, B, C, D, E, F, H, I, J, K, L, M, N: INV-assessed PFS per INRC | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: IRC-assessed Intracranial (IC)-ORR per RECIST v1.1 | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: IRC-assessed IC-DOR per RECIST v1.1 | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: IRC-assessed IC-CBR per RECIST v1.1 | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: IRC-assessed IC-PFS Rate per RECIST v1.1 | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: INV-assessed IC-ORR per RECIST v1.1 | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: INV-assessed IC-DOR per RECIST v1.1 | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: INV-assessed IC-CBR per RECIST v1.1 | Approximately up to 12 years
Cohorts A, B, C, D, I, J, K: INV-assessed IC-PFS Rate per RECIST v1.1 | Approximately up to 12 years
Cohorts A and B: Percentage of Participants With Confirmed Deterioration as Assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Approximately up to 12 years
  The EORTC QLQ-C30 is a validated, reliable self-report measure. It consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), eight symptom scales (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea) and global health/quality of life, with a recall period of the previous week. Scale scores can be obtained for the multi-item scales using rating scales of 4 or 7 points.
Cohorts A and B: Change From Baseline in the EORTC-QLQ-C30 Total Score | Approximately up to 12 years
  The EORTC QLQ-C30 is a validated, reliable self-report measure. It consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), eight symptom scales (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea) and global health/quality of life, with a recall period of the previous week. Scale scores can be obtained for the multi-item scales using rating scales of 4 or 7 points.
Cohorts A and B: Percentage of Participants With a Clinical Meaningful Change on the Global Health Status, Physical Functioning, and Role Functioning Scores From the EORTC QLQ-C30 | Approximately up to 12 years
  The EORTC QLQ-C30 is a validated, reliable self-report measure. It consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), eight symptom scales (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea) and global health/quality of life, with a recall period of the previous week. Scale scores can be obtained for the multi-item scales using rating scales of 4 or 7 points.
Cohorts A and B: Time to Confirmed Symptom Onset or Worsening From Tumor-related Symptom Scores From the EORTC QLQ-C30 and EORTC Item Library 71 (IL71) | Approximately up to 12 years
  The EORTC Item library includes stand-alone symptoms scales and an overall assessment of treatment bother to provide additional information not currently captured in the EORTC QLQ-C30. The scales use the same rating scale and recall period of previous week as the symptom scales in the EORTC QLQ-C30.
All Cohorts: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Approximately up to 12 years
  AE severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5 (NCI CTCAE v5.0.)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (162):
- United States (56):
  - Southern Cancer Center, Daphne, Alabama
  - Western Regional Medical Center at Cancer Treatment Centers of America, Goodyear, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - USC Norris Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - University of California at San Francisco, San Francisco, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Christiana Care Health Srvcs, Newark, Delaware
  - University of Florida, Gainesville, Florida
  - Miami Cancer Institute of Baptist Health, Inc., Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - St. Alphonsus, Boise, Idaho
  - Midwestern Regional Med Center, Zion, Illinois
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - New England Cancer Specialists, Scarborough, Maine
  - Maryland Hematology & Oncology. P.A., Silver Spring, Maryland
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Metro-Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Washington University, St Louis, Missouri
  - Intermountain Health St. Vincent Regional Hospital - Cancer Centers of Montana, Billings, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada - Eastern Avenue, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - National Translational Research Group, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Cancer and Blood Specialists - Setauket Medical Oncology, Port Jefferson Station, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - Barrett Cancer Center, Cincinnati, Ohio
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Consultants in Medical Oncology and Hematology, Broomall, Pennsylvania
  - Alliance Cancer Specialists, Horsham, Pennsylvania
  - Virginia Cancer Specialists - Leesburg, Leesburg, Pennsylvania
  - Cancer Treatment Centers of America, Philadelphia, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - PRISMA Health - Greenville, Greenville, South Carolina
  - The West Clinic, Germantown, Tennessee
  - St. Jude Children'S Research Hospital, Memphis, Tennessee
  - Texas Oncology - Central South, Austin, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Cook Childrens Medical Center, Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology- Northeast Texas, Tyler, Texas
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - Royal Darwin Hospital, Tiwi, Northern Territory
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Children's Hospital, Parkville, Victoria
- Belgium (5):
  - Cliniques Universitaires St-Luc, Brussels
  - GHdC Site Les Viviers, Charleroi
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Brazil (4):
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Hospital A. C. Camargo, São Paulo, São Paulo
  - Clínica Onco Star - Rede D'Or, São Paulo, São Paulo
- Canada (6):
  - BC Cancer ? Vancouver, Vancouver, British Columbia
  - London Health Sciences Centre · Victoria Hospital, London, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
- China (10):
  - Beijing Cancer Hospital, Beijing
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - Jilin Cancer Hospital, Changchun
  - West China Hospital - Sichuan University, Chengdu
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai East Hospital, Shanghai
  - Zhongshan Hospital Fudan Unvierstiy, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet, København Ø
- France (6):
  - Institut Bergonie, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital de la Timone, Marseille
  - Institut Universitaire du Cancer de Toulouse-Oncopole, Toulouse
  - Institut de Cancerologie Gustave-Roussy (IGR), Villejuif
- Germany (9):
  - Uniklinik Essen, Essen
  - Georg-August-Uniklinik, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf Onkologisches Zentrum Medizinische Klinik II, Hamburg
  - Medizinische Hochschule Zentrum Innere Medizin Abt.Gastroenterologie, Endokrinologie und Hepatologie, Hanover
  - SLK-Kliniken Heilbronn GmbH;Klinik für Innere Medizin III, Heilbronn
  - Praxis für Hämatologie, Onkologie und Palliativmedizin, Mönchengladbach
  - Klinikum der Universität München, Campus Großhadern, München
  - Universtitätsklinikum Ulm, Ulm
  - Uniklinikum, Comprehensive Cancer Center Mainfranken, Würzburg
- Hong Kong (2):
  - Hong Kong Children's Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Rabin MC, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky / Ichilov Hospital, Tel Aviv
- Italy (9):
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Ospedale Pediatrico Bambino Gesù - IRCCS, Rome, Lazio
  - Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Asst Degli Spedali Civili Di Brescia, Brescia, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Istituto Nazionale Tumori di Milano, Milan, Lombardy
  - Dipartimento di Scienze Pediatriche Adolescenza, Turin, Piedmont
  - Azienda Ospedaliera Meyer, Florence, Tuscany
  - Azienda Ospedaliera Universitaria Senese, U.O.C. Immunoterapia Oncologica, Siena, Tuscany
- Japan (3):
  - National Cancer Center Hospital East, Chiba
  - Kindai University Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
- Auckland City Hospital, Cancer and Blood Research, Auckland, New Zealand
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gda?sk
  - Narod.Inst.Onkol. im. M.Sklodowskiej - Curie-Panst.Inst.Bad, Warsaw
- IPO do Porto, Porto, Portugal
- PanOncology Trials, San Juan, Puerto Rico
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
- Medical Oncology Centre of Rosebank, Johannesburg, South Africa
- South Korea (7):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital- Adult Site, Seoul
  - Seoul National University Hospital- Pediatric Site, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center- Adult Site, Seoul
  - Samsung Medical Center- Pediatric Site, Seoul
- Spain (10):
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Clinica Universidad de Navarra Madrid, Madrid
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - START Madrid. Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario la Fe, Valencia
- Switzerland (4):
  - Universitätsspital Basel (USB), Basel
  - Ospedale Regionale di Bellinzona Medizin Onkologie, Bellinzona
  - Inselspital, Klinik und Poliklinik für Medizinische Onkologie, Bern
  - Unversitätsspital Zürich, Zurich
- Taiwan (5):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital-Linkou, Taoyuan
  - National Taiwan University Hospital, Zhongzheng Dist.
- United Kingdom (5):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - University College London Hospital, London
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Royal Manchester Children?s Hospital, Manchester
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Thomas DM, Kim JE, Barlesi F, Martens UM, Krzakowski M, Dziadziuszko R, Jeong JH, Daniele G, Wilson TR, Wu F, Simmons BP, Patel S, Sbirnac M, Kaul M, Gadgeel SM. TAPISTRY: A Phase II Study of Atezolizumab in Patients with Tumor Mutational Burden-High Tumors. Clin Cancer Res. 2026 Jan 9. doi: 10.1158/1078-0432.CCR-25-3336. Online ahead of print. PMID 41511400
- [Derived] Desai AV, Bagchi A, Armstrong AE, van Tilburg CM, Basu EM, Robinson GW, Wang H, Casanova M, Andre N, Campbell-Hewson Q, Wu Y, Cardenas A, Ci B, Ryklansky C, Devlin CE, Meneses-Lorente G, Wulff J, Hutchinson KE, Gajjar A, Fox E. Efficacy and safety of entrectinib in children with extracranial solid or central nervous system (CNS) tumours harbouring NTRK or ROS1 fusions. Eur J Cancer. 2025 May 2;220:115308. doi: 10.1016/j.ejca.2025.115308. Epub 2025 Feb 22. PMID 40086048